CLINICAL TRIAL: NCT06909942
Title: Association of Sarcopenia With Rocuronium Use in Liver Transplant Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, EMRE ARIKAN, Asisstant anesthesiologist, Inonu University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2025/7237
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Sarcopenia; Sarcopenia in Liver Cirrhosis; Liver Transplantation
Keywords: sarcopenia; psoas muscle index; handgrip dynamometer; liver transplantation
MeSH Terms: conditions — Sarcopenia | interventions — Neuromuscular Monitoring; Consciousness Monitors

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- liver transplantation recipients with sarcopenia (Active Comparator): this arm includes patient with sarcopenia in liver transplantation recipient group.They determined with SARC-F score , hangrip dynamometer value in kilogram and psoas muscle area measurement based on lomber CT scan .
  Interventions: Diagnostic Test: Psoas Muscle Index; Device: Handgrip Dynamometer; Other: SARC-F Score; Device: Train-of-Four(TOF); Device: Bispectral Index(BIS)
- liver transplantation recipients without sarcopenia (Placebo Comparator): the patients are this arm whom all going liver tranplantation for any reason but they have no sarcopenia in diagnosis algorithm
  Interventions: Diagnostic Test: Psoas Muscle Index; Device: Handgrip Dynamometer; Other: SARC-F Score; Device: Train-of-Four(TOF); Device: Bispectral Index(BIS)

INTERVENTIONS:
Diagnostic Test: Psoas Muscle Index — The PMI is typically calculated using cross-sectional imaging (CT or MRI) at the level of the third lumbar vertebra (L3).The total psoas area is normalized to patient height: PMI = Total psoas muscle area (cm²) / height² (m²).The PMI is particularly valuable in hospital settings where patients may have difficulty performing functional tests like handgrip strength measurements, offering an objective assessment of muscle status from readily available imaging data.
Device: Handgrip Dynamometer — Handgrip strength (HGS) is one of the key diagnostic criteria for sarcopenia according to several international consensus guidelines, including those from the European Working Group on Sarcopenia in Older People (EWGSOP2) and the Asian Working Group for Sarcopenia (AWGS).Men: <27 kg and women: <16 kg values indicates sarcopenia for each patient.Handgrip strength measurement with a dynamometer provides a standardized, reliable, and clinically relevant assessment that helps identify individuals with sarcopenia who may benefit from early intervention strategies.
Other: SARC-F Score — The SARC-F is a simple screening tool used to identify individuals at risk for sarcopenia, which is the progressive loss of muscle mass and strength typically associated with aging.
  The SARC-F questionnaire consists of 5 components that assess key aspects related to muscle function:
  Strength: Difficulty lifting and carrying 10 pounds Assistance with walking: Difficulty walking across a room Rising from a chair: Difficulty transferring from a chair or bed Climbing stairs: Difficulty climbing a flight of 10 stairs Falls: Frequency of falls in the past year
  Each component is scored from 0-2 points:
  0 = No difficulty
  1. = Some difficulty
  2. = A lot of difficulty or unable to do
  The total score ranges from 0-10, with higher scores indicating higher risk:
  A score of 4 or greater suggests risk of sarcopenia A score of less than 4 suggests low risk
Device: Train-of-Four(TOF) — A Train of Four (TOF) device is a specialized neuromuscular monitoring tool used primarily in anesthesiology and critical care to assess the degree of neuromuscular blockade in patients who have received neuromuscular blocking agents (NMBAs).The device delivers four sequential electrical stimuli (hence "train of four") at 0.5-second intervals to a peripheral nerve, typically the ulnar nerve at the wrist. It then measures the resulting muscle contractions, usually of the adductor pollicis muscle (thumb).Modern TOF devices provide a numerical value called the TOF ratio or count, which compares the strength of the fourth twitch to the first twitch.
  Ratio of fourth twitch to first twitch amplitude <0.7: Significant residual blockade 0.7-0.9: Moderate recovery 0.9: Adequate recovery for extubation
Device: Bispectral Index(BIS) — A Bispectral Index (BIS) device is a specialized monitoring system used primarily in anesthesiology and critical care to assess a patient's level of consciousness during sedation and general anesthesia.Uses a sensor placed on the patient's forehead to capture electroencephalogram (EEG) signals from the brain.Employs advanced algorithms to analyze the raw EEG data, examining frequency, power, and phase relationships.Processes the EEG information into a dimensionless number (the BIS value) ranging from 0 to 100.
  BIS Scale:
  100-80: Awake, normal consciousness 80-60: Light to moderate sedation 60-40: General anesthesia (surgical level of hypnosis) 40-20: Deep hypnotic state 20-0: Burst suppression to flatline EEG (very deep anesthesia)

SUMMARY:
Patients will be informed by obtaining consent when they meet the inclusion criteria.

Written consent will be obtained when the patient arrives in the operating room.

The patient's characteristics (gender, age, liver disease) and the biochemistry, hemogram and coagulation values taken before the surgery will be written on the prepared follow-up form.

After the hand grip strength is recorded in kg with a mechanical thenar muscle dynamometer, the SARC-F test questionnaire consisting of five questions will be administered to the patient and the SARC-F score will be calculated and recorded.

Routine monitoring (ECG, pulse oximetry, non-invasive blood pressure cuff, TOF monitoring, BIS monitoring) will be performed for the liver transplant recipient.

The routine anesthesia induction protocol will be applied to the patient for liver transplant recipients (thiopental (5-7 mg/kg), fentanyl (1-2 mcg/kg) and rocuronium (1mg /kg)), the time after rocuronium will be recorded and the reset time of the TOF device will be determined.

After intubation, the intubation score will be recorded on the follow-up form as a value between 5 and 20.

During the case, the times when the TOF value exceeds 30% and the times when diaphragm activity is detected at -3 cmH2O on mechanical ventilation will be recorded, 0.1 mg/kg rocuronium will be added as required for routine anesthesia follow-up. The phase of the transplant operation (Dissection-Anhepatic-Neohepatic) in which the added rocuronium is added will be specified.

The transfusion content and amounts within the case will be recorded on the follow-up form.

The extubation times in hours, the transfer time to the ward, the discharge time from the hospital and the need for reintubation of patients who are routinely transferred to the intensive care unit in an intubated state at the end of the case will be recorded.

DETAILED DESCRIPTION:
This prospective observational study will investigate the effect of sarcopenia on rocuronium use in patients scheduled for liver transplantation. The study population will consist of ASA II-III patients aged 18-65 years who are scheduled to undergo liver transplantation at İnönü University Liver Transplantation Institute. Sarcopenia assessment will be made with a three-stage algorithm: 1. SARC-F Questionnaire: A validated 5-question questionnaire evaluating muscle strength, walking aid, getting up from a chair, climbing stairs, and fall history will be applied. 2. Hand Grip Strength: Will be measured with a mechanical thenar muscle dynamometer and recorded in kg. Values will be compared with reference values determined according to gender. 3. Psoas Muscle Index (PMI): Psoas muscle area will be measured at the level of L3 vertebra on abdominal CT images taken preoperatively for the purpose of operation plan and liver volume evaluation. PMI will be calculated by dividing the total psoas muscle area (cm²) by the square of height (m²). PMI values will be classified according to cut-off values determined by gender. Patients will be informed by obtaining consent when they meet the inclusion criteria. Written consent will be obtained when the patient arrives in the operating room. The patient's characteristics (gender, age, liver disease) and the biochemistry, hemogram and coagulation values taken before the surgery will be written on the prepared follow-up form. After the hand grip strength is recorded in kg with a mechanical thenar muscle dynamometer, the SARC-F test questionnaire consisting of five questions will be applied to the patient and the SARC-F score will be calculated and recorded. Routine monitoring (ECG, pulse oximetry, non-invasive blood pressure cuff, TOF monitoring, BIS monitoring) will be performed for the liver transplant recipient. The patient will be administered the routine anesthesia induction protocol for liver transplant recipients (thiopental (5-7 mg/kg), fentanyl (1-2 mcg/kg) and rocuronium (1 mg/kg)), the time after rocuronium is administered will be recorded and the reset time of the TOF device, which is one of the routine anesthesia monitors, will be determined. After intubation, the intubation score will be written on the follow-up form as a value between 5 and 20. During the case, the times when the TOF value exceeds 30% and the times when diaphragm activity is detected at -3 cmH2O on the mechanical ventilator will be recorded, 0.1 mg/kg rocuronium will be added as required by routine anesthesia follow-up. The phase of the transplant operation (Dissection-Anhepatic-Neohepatic) in which the added rocuronium is added will be specified. The transfusion content and amounts in the case will be written on the follow-up form. The extubation times in hours, transfer times to the ward, discharge times from the hospital and the need for reintubation of patients who are routinely transferred to intensive care in an intubated state at the end of the case will be recorded in the postoperative process. Patients will be extubated using sugammadex, a direct rocuronium antagonist, routinely in the postoperative process.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists (ASA) 2-3,
* Patients over the age of 18,
* Liver transplant recipient candidates who have agreed to receive an organ transplant

Exclusion Criteria:

* Patients who are unconscious enough to not be included in the study (patients for whom consent cannot be obtained and the study cannot be explained)
* Patients under the age of 18
* Patients aged 65 and over
* Patients with advanced renal failure
* Patients with massive ascites in the abdomen
* Patients with advanced heart failure or high pulmonary artery pressure for whom routine anesthesia induction protocols must be excluded
* Patients with psychosis or substance abuse Patients with a known adverse reaction to rocuronium

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Idealising Rocuronium Dosing in Sarcopenic Patients With Using Sarcopenia Diagnostic Tests in Preoperative Period | From surgical prosedure to the end of ward observation at 6 months
  The dose of rocuronium is determined according to the body weight in kilograms of the patients in routine practice. The primary endpoint of our study is to determine whether sarcopenic patients can be identified and induction can be performed with a lower rocuronium dose(mg/kg) than the routine approach.

SECONDARY OUTCOMES:
It is aimed to reduce the length of stay of patients in the service and intensive care unit by adjusting the drug doses that will be used with the detection of sarcopenia | From surgical prosedure to the end of treatment at 6 months
  Postoperative residual neuromuscular blockade increases the risk of postoperative complications. The secondary endpoint of our study was to determine whether the possibility of residual blockade by using lower doses of rocuronium and identifying sarcopenic patients would reduce the duration of extubation time in hour, intensive care, and hospital stay(days).

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Altunkaya Yagci, asisst. prof., Study Director — Inonu University
Locations (1):
- Turgut Ozal Medicine Center Liver Transplantation Institute, Malatya, Battalgazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Takagi S, Sugaya N, Kiuchi N, Iwasa A, Itagaki M, Seki A, Suzuki J, Suzuki T. High-dose rocuronium-induced paralysis of the adductor pollicis muscle facilitates detection of the timing for tracheal intubation in elderly patients: a randomized double-blind study. J Anesth. 2020 Dec;34(6):876-880. doi: 10.1007/s00540-020-02831-6. Epub 2020 Jul 23. PMID 32705417
- [Result] Kuo SZ, Ahmad M, Dunn MA, Montano-Loza AJ, Carey EJ, Lin S, Moghe A, Chen HW, Ebadi M, Lai JC. Sarcopenia Predicts Post-transplant Mortality in Acutely Ill Men Undergoing Urgent Evaluation and Liver Transplantation. Transplantation. 2019 Nov;103(11):2312-2317. doi: 10.1097/TP.0000000000002741. PMID 30985575